CLINICAL TRIAL: NCT05077228
Title: Efficiency of the Imaging Strategy for the Management of Suspected Covid-19
Acronym: EFFI-COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7976
Record Dates: First submitted 2021-10-11; First posted 2021-10-14 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Dyspnea; Cough; Sputum; Diarrhea; Confusion
MeSH Terms: conditions — COVID-19; Dyspnea; Cough; Diarrhea; Confusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency departments have been placed at the heart of the patient triage strategy during the COVID-19 epidemic. In the absence of scientific knowledge on the most efficient strategy to put in place in emergency structures, the centers have proposed very heterogeneous protocols resulting from collaboration with local radiology and virology teams. While the pandemic in France appears to be currently under control, it is important to assess the sorting strategies put in place to deal with a new epidemic.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject treated in the emergency rooms of participating centers for suspicion of COVID-19 presenting with fever> 38 ° and / or respiratory signs (dyspnea, cough, sputum) and / or other symptoms suggestive of COVID-19 (diarrhea , confusion ...) and / or people over 85 or living in an institution during the study period from March 9 to May 8, 2020
* Subject affiliated to a social health insurance protection scheme
* Subject not having expressed their opposition, after information, to the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject treated in the emergency rooms of participating centers for suspicion of COVID-19 presenting with fever> 38 ° and / or respiratory signs (dyspnea, cough, sputum) and / or other symptoms suggestive of COVID-19 (diarrhea , confusion ...) and / or people over 85 or living in an institution during the study period from March 9 to May 8, 2020
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
A retrospective study of the imaging strategy for the management of suspected Covid-19 | Files analysed retrospectively from March 09, 2020 to May 08, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina GARNIER KEPKA, MD, Principal Investigator — Service d'accueil des urgences - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'accueil des urgences - Hôpitaux Universitaires de Strasbourg, Strasbourg, France